CLINICAL TRIAL: NCT06491849
Title: Observational Study on the Peri-implant/Screw Conditions of Mini Implants Placed During Orthodontic Treatment
Brief Title: Evaluation of Peri-implant Conditions of Orthodontic Mini Implants
Status: Completed | Type: Observational
Sponsor: Dr. Mehmet Selim Yildiz (Other)
Responsible Party: Sponsor-Investigator, Dr. Mehmet Selim Yildiz, Assistant Professor, Dr., Altinbas University
Organization: Altinbas University (Other)
Other Study IDs: 2021/49
Record Dates: First submitted 2024-06-28; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Dental Implantation; Peri-implant Mucositis; Gingival Inflammation; Implant Stability; Orthodontics
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthodontic Mini Implant Group: Participants with at least one orthodontic mini implant placed for anchorage during orthodontic treatment. The study will evaluate the peri-implant conditions, including gingival and mucosal inflammation, implant stability, and other related factors.
  Interventions: Other: Peri-implant Condition Evaluation

INTERVENTIONS:
Other: Peri-implant Condition Evaluation — This intervention involves a detailed clinical evaluation of peri-implant conditions in patients who have received orthodontic mini implants. The assessments include measuring periodontal parameters such as probing depth, bleeding on probing, mucosal redness, plaque index, gingival index, and implant stability. The evaluations are conducted at specified intervals during and after orthodontic anchorage treatment to monitor changes and ensure the health of peri-implant tissues.

SUMMARY:
This observational study aims to evaluate the peri-implant conditions of mini implants placed during orthodontic treatment. Orthodontic mini implants are commonly used as temporary anchorage devices to prevent or reduce unwanted tooth movements during orthodontic treatment. The stability of these implants, both primary and secondary, is crucial for their success. Primary stability refers to the mechanical locking between the implant and bone immediately after placement, while secondary stability is achieved through bone remodeling around the implant over time.

Factors affecting the stability and success of mini implants include the patient's age, gender, cortical bone thickness and density, the site of implant placement, the presence of mobile surrounding tissue, implant dimensions, surface characteristics, and the magnitude and duration of applied orthodontic forces. Peri-implantitis, an inflammation around the implant, is a significant risk factor for implant failure and is influenced by oral hygiene and the quality of surrounding soft tissue.

This study will observe and analyze the peri-implant conditions in patients receiving orthodontic treatment with mini implants, focusing on the incidence of gingival/mucosal inflammation and other factors that may affect implant stability and success.

DETAILED DESCRIPTION:
Study Title:

Evaluation of Peri-implant Conditions of Orthodontic Mini Implants

Objective:

The primary objective of this observational study is to evaluate the periodontal conditions surrounding orthodontic mini implants placed during orthodontic treatment. Additionally, the study aims to assess the impact of existing periodontal/peri-implant conditions on the stability of the mini implants.

Background:

Orthodontic mini screws/implants are commonly used as temporary anchorage devices to prevent or reduce unwanted tooth movements during orthodontic treatment. For these mini screws to function effectively as anchorage units, they must be resistant to the forces applied and remain stable at the site of placement throughout their use. Stability is classified into two types: primary stability, which is the mechanical locking between the implant and bone immediately after placement, and secondary stability, which results from bone remodeling around the implant over time. Both types of stability are crucial for the success of mini implants.

Several factors influence the stability and success of mini implants, including the patient's age, gender, cortical bone thickness and density, the site of implant placement, mobility of surrounding tissues, implant dimensions, surface characteristics, and the magnitude and duration of applied orthodontic forces. Peri-implantitis, an inflammation around the implant, is a significant risk factor for implant failure and is influenced by oral hygiene and the quality of surrounding soft tissues.

Hypothesis:

The hypothesis of this study is that the incidence of gingival/mucosal inflammation around the peri-implant/mini screw areas is high.

Methodology:

Patient Population:

The study will include patients treated at Altinbas University Dental Hospital's Departments of Periodontology and Orthodontics between March 2021 and March 2023. Patients must have at least one orthodontic mini implant placed and be systemically healthy. Patients with a history of prosthetic treatment or those taking medications that affect periodontal tissues (e.g., Cyclosporine-A, Calcium Channel Blockers, Phenytoin) will be excluded.

Clinical Assessments:

Primary Assessments:

Clinical periodontal/peri-implant measurements for the entire mouth and each mini implant/screw.

Bleeding on probing (yes/no), suppuration (yes/no), mucosal redness (erythema), plaque index (0-3), gingival index (0-3), probing depth (mm), clinical attachment loss (mm), width of keratinized mucosa (mm), peri-implant mucosal thickness (mm), and radiographic evaluation of the distance between the mini implant/screw and roots (mm).

Secondary Assessments:

Stability of the mini implants/screws measured using a torque gauge. Type of orthodontic force applied, method of placement (with or without a stent), surface characteristics, type (self-tapping/self-drilling), dimensions (diameter and length), duration of application, amount of force applied (<250 grams), and type of orthodontic force system (elastic/coil systems).

Statistical Analysis:

The study will utilize descriptive statistical methods to evaluate the collected data. Due to the original nature of the research, a power analysis could not be performed before the study.

Expected Outcomes:

The findings from this study are expected to highlight the importance of soft tissue health and maintenance during the planning, surgical placement, and post-operative phases of mini implant applications in orthodontics. Additionally, the study aims to elucidate the impact of existing oral hygiene on the stability and force continuity of mini implants in similar patient groups, thereby providing insights into the optimal frequency of periodontal maintenance for individuals with mini implant anchorage.

Study Location:

Altinbas University Dental Hospital, Zuhuratbaba Neighbourhood, Incirli St. No:11-A, 34147 Bakırköy, Istanbul, Turkey.

This detailed description provides a comprehensive overview of your study, outlining its objectives, background, methodology, and expected outcomes in a structured and academic manner.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have at least one orthodontic mini implant placed for anchorage during orthodontic treatment.
* Systemically healthy individuals.
* Participants without a history of prosthetic treatment.

Exclusion Criteria:

* Individuals taking medications that can affect periodontal tissues (e.g., Cyclosporine-A, Calcium Channel Blockers, Phenytoin).
* Individuals with a history of prosthetic treatment.
* Individuals without orthodontic mini implants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients who had been treated with orthodontic mini implants at the Department of Orthodontics, Faculty of Dentistry, Altinbas University. A total of 16 patients were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Gingival/Mucosal Inflammation | 3 months
  Measurement of gingival and mucosal inflammation around the orthodontic mini implants using clinical indices. Units of Measure:
  Gingival Index (GI) (0-3) Plaque Index (PI) (0-3)
Probing Pocket/Mucosal Depth | 3 months
  Measurement of the depth of periodontal pockets or mucosal depth around the mini implants. Unit of Measure: Millimeters (mm)
Clinical Attachment Loss (Gingival recession) | 3 months
  Measurement of the loss of attachment or gingival recession in the periodontal tissues and around the mini implants. Unit of Measure: Millimeters (mm)
Width of Keratinized Mucosa | 3 months
  Measurement of the width of keratinized mucosa around the mini implants. Unit of Measure: Millimeters (mm)
Thickness of Peri-Implant/Screw Mucosa | 3 months
  Measurement of the thickness of the mucosa around the mini implants. Unit of Measure: Thick/Thin
Radiographic Evaluation | 3 months
  Measurement of the distance between the mini implant/screw and adjacent roots. Unit of Measure: Millimeters (mm)
Bleeding on Probing | 3 months
  Assessment of the presence or absence of bleeding upon probing around the mini implants and teeth. Unit of Measure: Binary (Yes/No) and given as percentage by the site and full mouth.
Mucosal redness (Erythema) | 3 months
  Assessment of the presence and degree of mucosal redness around the mini implants.
  Unit of Measure: Binary (Yes/No)
Mucosal discomfort | 3 months
  Patient-reported discomfort in the area surrounding the mini implants. Unit of Measure: Binary (Yes/No)

SECONDARY OUTCOMES:
Implant Stability | 3 months
  Assessment of the stability of the orthodontic mini implants using a torque gauge to measure insertion and removal torque values. Unit of Measure: Torque (Ncm)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Selim Yildiz, Asst. Prof., Principal Investigator — Altinbas University, Faculty of Dentistry
Locations (1):
- Altinbas University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers can request access to the IPD by contacting Dr. Mehmet Selim Yildiz at "mehmet.yildiz2@altinbas.edu.tr"

REFERENCES:
- [Background] Ure DS, Oliver DR, Kim KB, Melo AC, Buschang PH. Stability changes of miniscrew implants over time. Angle Orthod. 2011 Nov;81(6):994-1000. doi: 10.2319/120810-711.1. Epub 2011 May 25. PMID 21612317
- [Background] Lee SJ, Ahn SJ, Lee JW, Kim SH, Kim TW. Survival analysis of orthodontic mini-implants. Am J Orthod Dentofacial Orthop. 2010 Feb;137(2):194-9. doi: 10.1016/j.ajodo.2008.03.031. PMID 20152674
- [Background] Samrit V, Kharbanda OP, Duggal R, Seith A, Malhotra V. Bone density and miniscrew stability in orthodontic patients. Aust Orthod J. 2012 Nov;28(2):204-12. PMID 23304969
- [Background] Zitzmann NU, Berglundh T, Ericsson I, Lindhe J. Spontaneous progression of experimentally induced periimplantitis. J Clin Periodontol. 2004 Oct;31(10):845-9. doi: 10.1111/j.1600-051X.2004.00567.x. PMID 15367187
- [Background] Park HS, Jeong SH, Kwon OW. Factors affecting the clinical success of screw implants used as orthodontic anchorage. Am J Orthod Dentofacial Orthop. 2006 Jul;130(1):18-25. doi: 10.1016/j.ajodo.2004.11.032. PMID 16849067
- [Background] Parmar R, Reddy V, Reddy SK, Reddy D. Determination of soft tissue thickness at orthodontic miniscrew placement sites using ultrasonography for customizing screw selection. Am J Orthod Dentofacial Orthop. 2016 Oct;150(4):651-658. doi: 10.1016/j.ajodo.2016.03.026. PMID 27692423
- [Derived] Yildiz MS, Ulutas PA, Ozenci I, Akcali A. Clinical and radiographic assessment of the association between orthodontic mini-screws and periodontal health. BMC Oral Health. 2024 Nov 14;24(1):1376. doi: 10.1186/s12903-024-05136-2. PMID 39543578